CLINICAL TRIAL: NCT00749723
Title: Therapy-Optimization Trial and Phase II Study for the Treatment of Relapsed or Refractory of Primitive Neuroectodermal Brain Tumors and Ependymomas in Children and Adolescents
Brief Title: Therapy Optimization Trial for the Treatment of Relapsed or Refractory Brain Tumors in Children
Acronym: HIT-REZ-2005
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Gudrun Fleischhack, MD, Department of Pediatric Hematology & Oncology, Pediatrics III, University Children's Hospital Essen, University Hospital, Essen
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2005-002618-40; BfArM-4030755 (Other: Federal Institute for Drugs and Medical Devices (BfArM)); EC-105/05 (Other: Leading Ethic Committee University Hospital of Bonn); DKS 2006.01, 2008.17, 2012.03 (Other Grant/Funding Number: German Children Cancer Foundation)
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Brain Tumors; Supratentorial PNETs; Medulloblastomas; Ependymomas
Keywords: brain tumor; relapse; children; etoposide; intraventricular; temozolomide
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma; Ependymoma; Recurrence | interventions — Carboplatin; Etoposide; Temozolomide; Thiotepa; trofosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1: P-HIT-REZ 2005 (Experimental): intravenous chemotherapy with carboplatin/etoposide,followed by
  * high dose chemotherapy with thiotepa, carboplatin, etoposide and autologous stem cell transplantation if patient have achieved a complete remission or
  * maintenance therapy with oral trofosfamide, etoposide
  Interventions: Drug: carboplatin; Drug: etoposide; Drug: thiotepa, carboplatin, etoposide; Procedure: autologous stem cell transplantation; Drug: intraventricular etoposide; Drug: trofosfamide, etoposide
- 2: P-HIT-REZ 2005 (Experimental): oral chemotherapy with temozolomide, followed by
  * high dose chemotherapy with temozolomide, thiotepa and autologous stem cell transplantation if patient have achieved a complete remission
  * maintenance therapy with oral temozolomide or in case of progression with oral trofosfamide, etoposide
  Interventions: Drug: temozolomide; Drug: temozolomide, thiotepa; Procedure: autologous stem cell transplantation; Drug: intraventricular etoposide
- 3: E-HIT-REZ 2005 (Experimental): Phase II: oral chemotherapy with temozolomide after progression oral trofosfamide, etoposide
  Interventions: Drug: temozolomide; Drug: intraventricular etoposide; Drug: trofosfamide, etoposide
- Intraventricular Etoposide (Experimental): Phase II, intraventricular chemotherapy with etoposide
  Interventions: Drug: intraventricular etoposide

INTERVENTIONS:
Drug: carboplatin — 200 mg/m²/d continuously IV on day 1-4 of each 21-28-day-cycle. Number of cycles: until disease progression, maximum 4 cycles
  Other Names: Carboplatin IV
  Arms: 1: P-HIT-REZ 2005
Drug: etoposide — 100mg/m²/d continuously IV on day 1-4 of each 21-28 day cycle. Number of cycles: until disease progression, maximum 4 cycles
  Other Names: etoposide IV
  Arms: 1: P-HIT-REZ 2005
Drug: temozolomide — 150mg/m²/d p.o. on day 1-5 of a 21-28-day-cycle. Number of cycles: until progression or maximum up to 2 years
  Other Names: temozolomide orally
  Arms: 2: P-HIT-REZ 2005; 3: E-HIT-REZ 2005
Drug: thiotepa, carboplatin, etoposide — high dose chemotherapy followed by to autologous stem cell transplantation
  Other Names: thiotepa, carboplatin, etoposide IV, high dose
  Arms: 1: P-HIT-REZ 2005
Drug: temozolomide, thiotepa — high dose chemotherapy followed by autologous stem cell transplantation
  Other Names: temozolomide, thiotepa IV
  Arms: 2: P-HIT-REZ 2005
Procedure: autologous stem cell transplantation — autologous stem cell transplantation following HD-chemotherapy
  Other Names: ASCT
  Arms: 1: P-HIT-REZ 2005; 2: P-HIT-REZ 2005
Drug: intraventricular etoposide — prior to systemic chemotherapy as single agent in patients with neoplastic meningitis, in addition to systemic chemotherapy if proven effective in phase II study, intraventricularly age-dependent daily dose (>3m to <3y 0.7 mg; >3y 1.0 mg) for 5 days every 2 two 4 weeks. Number of cycles: at least 3 courses, maximum up to 2 years
  Other Names: etoposide intra-CSF
Drug: trofosfamide, etoposide — maintenance therapy: trofosfamide and etoposide: 100 mg/m²/d and 25 mg/m²/d, respectively, for 21 days every 4 weeks. Number of cycles: until progression or maximum up to 2 years
  Other Names: trofosfamide, etoposide orally
  Arms: 1: P-HIT-REZ 2005; 3: E-HIT-REZ 2005

SUMMARY:
The purpose of this study is to improve overall survival while maintaining a good quality of life in pediatric patients with refractory or recurrent brain tumors (medulloblastomas, supratentorial PNETs, ependymomas WHO grade II and III). Response to different chemotherapy options (intravenous versus oral chemotherapy, intraventricular chemotherapy) as part of a multimodal therapy will be assessed. Progression-free, overall survival and toxicity will be evaluated additionally.

DETAILED DESCRIPTION:
Parts of the study:

P-HIT-REZ-2005: a trial for the treatment of relapsed PNETs (medulloblastomas,supratentorial PNETs)

E-HIT-REZ-2005: a trial for the treatment of relapsed ependymomas (Phase II-Study with temozolomide)

Phase II-Study: intraventricular therapy with etoposide in neoplastic meningitis in relapsed PNETs and ependymomas with subarachnoid tumor manifestation (window study)

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics

* Histologically confirmed Medulloblastoma, cerebral PNET or Ependymoma
* Refractory or relapsed disease
* Measurable disease by MRI or detection of tumor cells in cerebrospinal fluid Patients characteristics
* Performance status ECOG ≥ 3 or Karnofsky Status ≥ 40%
* Life expectancy ≥ 8 weeks

Hematological:

* Absolute leukocyte count ≥ 2.0 x 10^9 /l
* Hemoglobin ≥ 10g/dl
* Platelet count ≥ 70 x 10^9/l

Renal:

* Creatinine no greater than 1.5 times UNL
* No overt renal disease

Hepatic:

* Bilirubin less than 2.5 times UNL
* AST and ALT less than 5 times UNL
* No overt hepatic disease

Pulmonary:

* No overt pulmonary disease

Cardiovascular:

* No overt cardiovascular disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection Prior concurrent therapy
* More than 2 weeks since prior systemic chemotherapy
* More than 4 weeks since prior radiotherapy
* No other concurrent anticancer or experimental drugs Examinations required
* Examination of lumbar CSF
* Cranial and spinal MRI within 14 days prior to start of treatment

Ages: 3 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 174 (Actual)
Dates: Start 2006-02-01; Primary Completion 2015-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
P-HIT-REZ 2005 study: two Chemotherapy-arms: response evaluation after the fourth therapy course | 4 months for each patient (8 years for the whole study population)
  determination of objective repsonse rate (CR+PR)
E-HIT-REZ 2005 study (Phase II Study "Oral chemotherapy with temozolomide"): Evaluation of response rate to the 60-days oral chemotherapy with temozolomide | 2 months for each patient (8 years for the whole study population)
  determination of objective repsonse rate (CR+PR/all patients)
Phase II study "Intraventricular therapy with etoposide": Evaluation of response rate to the 5-week intraventricular therapy with etoposide | 6 weeks for each patient (8 years for the whole study population)
  disease stabilization rate (CR+PR+SD/all patients)

SECONDARY OUTCOMES:
P-HIT-REZ 2005 study: two Chemotherapy-arms: PFS and OS from start of therapy | 10 years
  progression free and overall survival from start of therapy until PD, last follow up or death, respectively
P-HIT-REZ 2005 study: two Chemotherapy-arms: toxicity rate (CTC) in both arms | 8 years
  rate of adverse events of CTC°3 or CTC°4 according to CTCAE v3.0
E-HIT-REZ 2005 study: Chemotherapy-arm: PFS and OS from start of therapy | 10 years
  progression free and overall survival from start of therapy until PD, last follow up or death, respectively
E-HIT-REZ 2005 study: Chemotherapy-arm: toxicity rate (CTC) | 10 years
  progression free and overall survival from start of therapy until PD, last follow up or death, respectively
Phase II study "Intraventricular therapy with etoposide": toxicity rate (CTC) | 8 years
  rate of adverse events of CTC°1-4 according to CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Gudrun Fleischhack, MD, Principal Investigator — Department of Pediatric Hematology & Oncology, Pediatrics III, University Children's Hospital Essen
Locations (54):
- Germany (54):
  - Universitätskinderklinik Aachen, Aachen
  - Klinikum Augsburg, Klinik für Kinder- und Jugendmedizin, Augsburg
  - Helios Klinikum Berlin-Buch, Klinik für Kinderheilkunde und Jugendmedizin, Berlin
  - Charité Klinikum Campus Virchow, Kinderklinik, Berlin
  - Klinik ür Kinder- und Jugendmedizin in Bethel, Bielefeld
  - Universitätskinderklinik Bonn, Bonn
  - Städtisches Klinikum Braunschweig, Kinderklinik, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Universitätskinderklinik Köln, Cologne
  - Carl-Thiele-Klinikum Cottbus, Zentrum für Kinderheilkunde, Cottbus
  - Vestische Kinder- und Jugendklinik Datteln, Datteln
  - Klinikum Dortmund, Klinik für Kinder- und Jugendmedizin, Dortmund
  - Universitätsklinikum Dresden, Kinderklinik, Dresden
  - Klinikum Duisburg, Klinik für Kinder-und Jugendmedizin, Duisburg
  - Universitätskinderklinik Düsseldorf, Düsseldorf
  - Helios Klinikum Erfurt, Zentrum für Kinderheilkunde, Erfurt
  - Universitätskinderklinik Erlangen, Erlangen
  - Universitätskinderklinik Essen, Essen
  - Klinikum der Wolfgang Goethe Universität, Klinik für Kinderheilkunde, Frankfurt am Main
  - Universitätskinderklinik Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg, Zentrum für Kinderheilkunde, Giessen
  - Universitätskinderklinik Göttingen, Göttingen
  - Universitätskinderklinik Greifswald, Greifswald
  - Martin-Luther-Universität Halle Wittenberg, Halle
  - Universitätskinderklinik Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule, Zentrum für Kinderheilkunde, Hanover
  - Universitätskinderklinik Heidelberg, Heidelberg
  - SLK Kinderklinik Heilbronn, Heilbronn
  - Gemeinschaftskrankenhaus Herdecke, Kinderklinik, Herdecke
  - Universitätskinderklinik, Homburg/Saar
  - Friedrich Schiller Universität, Klinik für Kinder-und Jugendmedizin, Jena
  - Städtisches Krankenhaus, Klinik für Kinder- und Jugendmedizin, Karlsruhe
  - Klinikum Kassel, Kinderklinik, Kassel
  - UKSH, Campus Kiel, Klinik für Allg. Pädiatrie, Kiel
  - Städtisches Klinikum Kemperhof, Klinik für Kinder- und Jugendmedizin, Koblenz
  - Universitätskinderklinik Leipzig, Leipzig
  - Universitätskinderklinik Lübeck, Lübeck
  - Otto-von-Guericke-Universität, Zentrum für Kinderheilkunde, Magdeburg
  - Universitätskinderklinik Mainz, Mainz
  - Universitätskinderklinik Mannheim, Mannheim
  - Universitätskinderklinik Marburg, Marburg
  - Klinikum Minden III, Klinik für Kinder-und Jugendheilkunde, Minden
  - Dr. von Haunersches Kinderspital, München
  - Städtisches Krankenhaus München-Schwabing, Kinderklinik der TU München, München
  - Universitätskinderklinik Münster, Münster
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinikum Oldenburg, Zentrum für Kinder-und Jugendmedizin, Oldenburg
  - Universitäts-Kinderklinik, Regensburg
  - Universitätskinderklinik Rostock, Rostock
  - Asklepios Klinik Sankt Augustin GmbH, Sankt Augustin
  - Olgahospital-Pädiatrisches Zentrum, Stuttgart
  - Universitätskinderklinik Tübingen, Tübingen
  - Univeritätsklinikum Ulm, Abteilung Kinder-und Jugendmedizin, Ulm
  - Universitätskinderklinik Würzburg, Würzburg

REFERENCES:
- See also: German Society of Pediatric Hematology and Oncology — http://www.kinderkrebsinfo.de/
- See also: German Children's Cancer Foundation — http://www.kinderkrebsstiftung.de/